CLINICAL TRIAL: NCT01952535
Title: A Randomized, Double-blind, Placebo-controlled Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Study of Administrating Single Ascending Dose of HMS5552 in Healthy Adult Volunteers
Brief Title: A Clinical Study to Evaluate Safety, Tolerability and Pharmacokinetics of Oral HMS5552 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hua Medicine Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMM0101
Record Dates: First submitted 2013-09-22; First posted 2013-09-30 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dorzagliatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- HMS5552 dose 1 (Experimental): A single dose of HMS5552 tablets (5~50mg) taken orally.
  Interventions: Drug: HMS5552; Drug: Placebo
- HMS5552 dose 2 (Experimental): A single dose of HMS5552 tablets (5~50mg) taken orally.
  Interventions: Drug: HMS5552; Drug: Placebo
- HMS5552 dose 3 (Experimental): A single dose of HMS5552 tablets (5~50mg) taken orally.
  Interventions: Drug: HMS5552; Drug: Placebo
- HMS5552 dose 4 (Experimental): A single dose of HMS5552 tablets (5~50mg) taken orally.
  Interventions: Drug: HMS5552; Drug: Placebo
- HMS5552 dose 5 (Experimental): A single dose of HMS5552 tablets (5~50mg) taken orally.
  Interventions: Drug: HMS5552; Drug: Placebo
- HMS5552 dose 6 (Experimental): A single dose of HMS5552 tablets (5~50mg) taken orally.
  Interventions: Drug: HMS5552; Drug: Placebo

INTERVENTIONS:
Drug: HMS5552
Drug: Placebo

SUMMARY:
The objectives of this study is to determine the safety profiles, tolerability, pharmacokinetics and pharmacodynamics of HMS5552 following single ascending doses in healthy adult subjects.

DETAILED DESCRIPTION:
This will be a randomized, double-blind and placebo-controlled safety study with single oral doses of HMS5552 given to healthy volunteers.

The primary objective is to characterize the safety profiles of HMS5552 following single ascending doses (SAD) in healthy adult subjects.

The secondary objectives include:

1. To assess the pharmacokinetic profiles of HMS5552 after single dosing
2. To assess the preliminary pharmacodynamic profiles of HMS5552

Each study subject will receive a single oral dose of HMS5552. During each dosing, eight subjects will be allocated to receive HMS5552 and two subjects will be allocated to receive placebo treatment.

Several doses of HMS5552 will be tested. Dose titration or reduction is determined for each cohort based on the safety and pharmacokinetic data obtained from the lower dose cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Female and male volunteers, 18 to 45 years of age
* BMI: 18 to 24 kg/m2
* Fasting plasma glucose: 3.9 to 6.1 mmol/L
* Glucose level at 2 hours following oral glucose tolerance test <7.8 mmol/L
* HbA1c: 4 to 6.5%
* Normal supine blood pressure and normal ECG recordings

Exclusion Criteria:

* Female with child-bearing potential
* Evidence of clinically-significant renal, cardiac, bronchopulmonary, vascular, gastrointestinal, allergic, neurologic, metabolic (diabetes, thyroid disorders, adrenal disease), immunodeficiency disorders, cancer, hepatitis or cirrhosis.
* Intake of grapefruit or anything that may affect liver enzyme function within 1 month prior to the dosing day
* Clinically-relevant deviation from normal in the physical examination
* Subjects with a medical disorder, condition or history of such that would impair the subject's ability to participate or complete this study in the opinion of the investigator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of HMS5552 will be assessed by adverse event monitoring, physical examinations, 12 lead ECGs, vital sign, and safety laboratory measurements. | up to 72 hours post-dose

SECONDARY OUTCOMES:
The single dose pharmacokinetics of HMS5552 will be described by estimating parameters of AUCinf, AUC0-t, Cmax, Tmax, Ae, T1/2. | up to 72 hours post-dose
  Plasma will be collected at predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hour post-dose. Urine will be collected at predose, 0 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48, and 48 to 72 hour post-dose.
Pharmacodynamic variables will include maximum change (%) in fasting plasma glucose level, AUC0-4 of fasting plasma glucose , AUC of percent reduction in fasting plasma glucose from baseline versus time curve, time of minimum glucose level | up to 6 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: XueNing LI, MD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Hua Medicine Limited, Shanghai, Shanghai Municipality, China